CLINICAL TRIAL: NCT01731301
Title: A Pilot Study to Treat Patients With Chronic HCV Genotype 1 and ESRD Receiving Hemodialysis and Naïve to Prior HCV Therapy With Peginterferon Alfa-2b, the Maximally Tolerated Ribavirin Dose and Boceprevir
Brief Title: A Pilot Study to Treat Patients With Chronic Hepatitis C Virus (HCV) Genotype 1 and End-Stage Renal Disease (ESRD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liver Institute of Virginia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Chronic Liver Disease Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIV01
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Hepatitis C; End Stage Renal Disease
Keywords: Chronic hepatitis C; HCV; End stage renal disease; ESRD; Boceprevir; Ribavirin; Peg-interferon; Triple therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Kidney Failure, Chronic | interventions — Ribavirin; peginterferon alfa-2b; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ribavirin, peginterferon, boceprevir (Experimental): The efficacy and safety of HCV treatment in patients with ESRD will be assessed with a maximal tolerated dose of ribavirin, peginterferon and boceprevir.
  Interventions: Drug: Ribavirin; Drug: Peginterferon; Drug: Boceprevir

INTERVENTIONS:
Drug: Ribavirin — Ribavirin monotherapy will be started at a dose of 100 mg daily. After each successive week the dose of ribavirin will be increased by 100 mg increments daily as long as the hemoglobin remains greater than 10 gm/dl and/or there has not been a decline in the hemoglobin by more than 2 gms/dl from the pretreatment baseline.
  Other Names: Rebetol
Drug: Peginterferon — After the patient has remained on their maximal tolerated dose of ribavirin for 1 week peginterferon alpha-2b will be initiated at a dose of 1.0 mcg/kg/week. This dose was chosen because it is known to be equivalent in achieving SVR when compared to the 1.5 mcg/kg/dose and is associated with less bone marrow suppression. The dose of ribavirin will be adjusted as needed.
  Other Names: PegIntron, Rebetol and Victrelis
Drug: Boceprevir — Boceprevir will be added after the patient is on stable doses of ribavirin and peginterferon. The dose of ribavirin will be adjusted as needed.
  Other Names: Victralis

SUMMARY:
1. A maximally tolerated dose of ribavirin can be defined in each patient with ESRD undergoing hemodialysis.
2. Patients with Chronic Hepatitis C Virus (HCV)and End-Stage Renal Disease (ESRD)undergoing hemodialysis will be able to tolerate and remain on treatment with peginterferon alfa-2b, the maximally tolerated dose of ribavirin and boceprevir.
3. A significant percentage of patients with chronic HCV and ESRD undergoing hemodialysis can achieve rapid virologic response (RVR), extended virologic response (eRVR) and sustained virologic response (SVR) when treated with peginterferon alfa-2b, the maximally tolerated dose of ribavirin and boceprevir.

DETAILED DESCRIPTION:
Patients with ESRD will be treated with a dose escalation of ribavirin starting from 200 mg everyday (QD) to a maximal tolerated dose. Peginterferon will then be added. Ribavirin will be dose adjusted as needed. Boceprevir will then be added. Ribavirin will be dose adjusted as needed. Patients will be monitored for eRVR and SVR. The study end-point is eRVR.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV defined by:
* A history of a positive anti-HCV or HCV RNA for > 6 months or
* A liver biopsy demonstrating at least portal fibrosis
* HCV genotype 1
* No prior treatment with any interferon or peginterferon preparation
* ESRD undergoing hemodialysis for at least 6 months
* Willingness not to conceive a child during treatment and for 6 months following discontinuation of treatment.

Exclusion Criteria:

* Histologic evidence of cirrhosis
* Any co-existent liver disease
* A platelet count < 90,000
* A total white blood cell (WBC) < 2.5
* An absolute neutrophil count < 1.5
* Hemoglobin < 11 gm/dl on Epoetin-alpha
* Positive test for anti-HIV
* Pregnancy of the patient or their intimate partner
* Women who are breast feeding
* Significant cardiovascular disease
* History of suicide intent, severe depression requiring hospitalization or significant psychiatric disease
* Malignancy within 5 years of enrollment except for squamous or basal cell skin cancer
* Co-existent immune disorder such as lupus, rheumatoid as arthritis, colitis, Crohns disease, sarcoidosis, etc.
* Any patient in the opinion of the investigator who would not be a satisfactory study candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who achieve eRVR at treatment week 28 | 28 weeks
  The primary end-point for evaluation will be the percentage of patients who achieve eRVR at treatment week 28.

SECONDARY OUTCOMES:
Tolerability of treatment | 48 weeks
  A. The ability to define the maximal tolerated dose of ribavirin. B. The ability to remain on peg-interferon alfa-2b, ribavirin and boceprevir for 24 weeks C. The percentage of patients who achieve SVR

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell L Shiffman, MD, Principal Investigator — Liver Institute of Virginia, Bon Secours Health System
Locations (1):
- Liver Institute of Virginia, Richmond, Virginia, United States